CLINICAL TRIAL: NCT04632979
Title: Backward Running on a Negative Slope as a Treatment for Achilles Tendinopathy in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meuhedet. Healthcare Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MeuhedetHCO1
Record Dates: First submitted 2020-11-09; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2019-09

CONDITIONS: Achilles Tendinopathy
Keywords: Achilles tendinopathy; backward running; exercise; running overuse injury
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Backward runners (Experimental): Training protocol patients
  Interventions: Procedure: Backwards running on a Treadmil with a negative slope

INTERVENTIONS:
Procedure: Backwards running on a Treadmil with a negative slope — Running backward on a treadmill with a negative slope

SUMMARY:
This study will look to evaluate the feasibility of a backwards downhill running program as an option for the treatment of Achilles tendinopathy in runners. It is known that exercise on the Achilles tendon during elongation (eccentric exercise) improves tendon function after injury. However, during recovery, the patient is required to stop tendon-loading activities such as jumps and sprints. Therefore, during recovery, athletes decline in physical fitness.

Backward running on a negative slope can achieve a biomechanical load similar to eccentric exercise without decreasing physical fitness.

DETAILED DESCRIPTION:
The study was a prospective, single-arm feasibility study. Participants were patients who met the entry criteria and were referred to the Meuhedet health service Physical Therapy outpatient clinic, Jerusalem, from September 2019 to February 2020. The sample size was based on previous recommendations for pilot and feasibility studies (Julious 2005; Billingham, Whitehead, and Julious 2013). Inclusion criteria were: AT that was clinically determined by an orthopedic surgeon (E.S) according to nontraumatic pain and tenderness at the Achilles tendon and report of decreased activity levels secondary to Achilles pain; a history of running for at least one session a week in the past three months; age > 18 and < 70. Exclusion criteria were having other lower extremity injuries; prior treatment with eccentric exercise or currently receiving Physical Therapy for AT; received a steroid injection into the tendon in the three months prior, or underwent Achilles tendon surgery.

Participants received a total of nine treatment sessions, twice a week for a total of five weeks. Each treatment consisted of backward walking / running over an 8º negatively inclined treadmill. (Landice L7 Rehabilitation treadmill, New Jersey, USA) with a warmup and a cooldown on a stationary bike. A detailed description of the protocol is presented in Table 1. As backward locomotion on a treadmill was novel for all participants they were advised to hold the treadmill handles during the adjustment period (treatment sessions 1-3). Participants were also instructed to refrain from specific sports which involve continuous jumping and forward running throughout the intervention period. Patients were informed that if they do not feel comfortable with the training protocol, they could terminate their participation at any point.

Assessments took place at baseline, pretreatment four, pretreatment six, and at a separate meeting after treatment nine

ELIGIBILITY:
Inclusion Criteria:

1. Distinct tenderness of Achilles tendon with no pain in the neighboring structures.
2. Nontraumatic diffuse pain in the posterior calf with local tenderness in the Achilles tendon.
3. A history of running for at least one session a week in the past three months.
4. Age > 18 and < 70

Exclusion Criteria:

1. Achilles pain longer than six months.
2. Patients with an additional lower extremity injury unable to bear full weight on the limb.
3. Patients who are currently receiving physical therapy for Achilles tendinopathy, have received a steroid injection into the tendon in the three months prior, or underwent Achilles tendon surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
VISA-A questionnaire | baseline
  Subjective questionnaire specific for Achilles tendinopathy
VISA-A questionnaire | two weeks
  Subjective questionnaire specific for Achilles tendinopathy
VISA-A questionnaire | three weeks
  Subjective questionnaire specific for Achilles tendinopathy
VISA-A questionnaire | five weeks
  Subjective questionnaire specific for Achilles tendinopathy
Number of single legged heel raises from a flat surface before the onset of pain | baseline
  Heel raise height will be defined by a pretest of one maximum single legged heel raise assessed by a measuring tape in centimeters
Number of single legged heel raises from a flat surface before the onset of pain | two weeks
  Heel raise height will be defined by a pretest of one maximum single legged heel raise assessed by a measuring tape in centimeters
Number of single legged heel raises from a flat surface before the onset of pain | three weeks
  Heel raise height will be defined by a pretest of one maximum single legged heel raise assessed by a measuring tape in centimeters
Number of single legged heel raises from a flat surface before the onset of pain | five weeks
  Heel raise height will be defined by a pretest of one maximum single legged heel raise assessed by a measuring tape in centimeters
Onset of relevant Achilles tendon pain (measured in seconds) during Forward running at a self-selected comfortable pace on a treadmill | baseline
  Forward running on treadmill until the onset of relevant pain
Onset of relevant Achilles tendon pain (measured in seconds) during Forward running at a self-selected comfortable pace on a treadmill | three weeks
  Forward running on treadmill until the onset of relevant pain
Onset of relevant Achilles tendon pain (measured in seconds) during Forward running at a self-selected comfortable pace on a treadmill | five weeks
  Forward running on treadmill until the onset of relevant pain
Compliance | five weeks
  Treatment sessions will be calculated upon the patient's completion of the full treatment protocol for that specific session. Inclusion will be terminated upon lack of fulfilling the treatment protocol or failing to complete a total of at least eight sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Springer, prof, Study Director — Ariel University, Physical Therapy Department
Locations (1):
- Meuhedet Health Services, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braunstein M, Baumbach SF, Herterich V, Bocker W, Polzer H. [Acute achilles tendon rupture : State of the art]. Unfallchirurg. 2017 Dec;120(12):1007-1014. doi: 10.1007/s00113-017-0420-4. German. PMID 29038897
- [Background] Bovend'Eerdt TJ, Botell RE, Wade DT. Writing SMART rehabilitation goals and achieving goal attainment scaling: a practical guide. Clin Rehabil. 2009 Apr;23(4):352-61. doi: 10.1177/0269215508101741. Epub 2009 Feb 23. PMID 19237435
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782